CLINICAL TRIAL: NCT03385720
Title: Submandibular Gland Preservation During Neck Dissection for Oral Squamous Cell Carcinoma
Brief Title: Submandibular Gland Preservation in Neck Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang-Yan Yu (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Peking University School of Stomatology (Unknown)
Responsible Party: Sponsor-Investigator, Guang-Yan Yu, President of Chinese Stomatological Association, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sujiazeng
Record Dates: First submitted 2017-12-06; First posted 2017-12-28 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Neck Dislocation; Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Procedure: modified neck dissection
- Control group (Active Comparator)
  Interventions: Procedure: traditional neck dissection

INTERVENTIONS:
Procedure: modified neck dissection — Modified neck dissection with preservation of submandibular gland. The submandibular gland is preserved during neck dissection.
  Arms: Experimental group
Procedure: traditional neck dissection — traditional neck dissection without preservation of submandibular gland
  Arms: Control group

SUMMARY:
Trial design: a randomized controlled trial.

Eligibility criteria for participants: patients with primary early stage oral squamous cell carcinoma. Exclusion criteria: cancer of the floor of the mouth.

Interventions: submandibular gland is preserved during neck dissection for patients of the experimental group; submandibular gland is removed during neck dissection for patients of the control group.

Primary Parameters: survival rate, mortality rate

ELIGIBILITY:
Inclusion Criteria:

Primary oral squamous cell carcinoma of early stage (T1N0 and T2N0).

Exclusion Criteria:

Cancer of the floor of the mouth.

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
5-year survival rate | 5-year after operation
  disease free survival rate
3-year survival rate | 3-year after operation
  disease free survival rate
5-year regional recurrence rate | 5-year after operation
  rate of participants with tumor recurrence in the neck
3-year regional recurrence rate | 3-year after operation
  rate of participants with tumor recurrence in the neck
1-year regional recurrence rate | 1-year after operation
  rate of participants with tumor recurrence in the neck

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University School of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No